CLINICAL TRIAL: NCT01594216
Title: A Phase II Trial Of The JAK-Inhibitor Ruxolitinib (INCB018424) In Combination With Exemestane For Patients With Estrogen Receptor (ER) Positive Advanced Breast Cancer)
Brief Title: Ruxolitinib in Estrogen Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02112
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Estrogen-receptor Positive Invasive Metastatic Breast Cancer
Keywords: Postmenopausal female
MeSH Terms: interventions — ruxolitinib; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First Stage (Experimental): Ruxolitinib at 25 mg orally, twice daily and Exemestane, 25 mg orally once daily
  Interventions: Drug: Ruxolitinib; Drug: Exemestane
- Second Stage (Experimental): Ruxolitinib at 15 mg orally, twice daily and Exemestane, 25 mg orally once daily
  Interventions: Drug: Ruxolitinib; Drug: Exemestane

INTERVENTIONS:
Drug: Ruxolitinib
Drug: Exemestane

SUMMARY:
This is a Phase II investigator-Initiated trial of the Investigational Drug, Ruxolitinib, in combination with Exemestane in patients with estrogen-receptor positive advanced breast cancer. The objective of this study is to determine the preliminary safety and efficacy of the combination of exemestane and Ruxolitinib (INCB018424).

DETAILED DESCRIPTION:
In vitro mechanisms link IL-6 to poor outcome in breast cancer via activated JAK/STAT tumor signaling, leading to an aggressive tumor phenotype, and our preliminary data support these mechanisms in women with ER+ disease. Our overarching hypotheses are that (1) IL-6 mediates upregulation of JAK/STAT signaling pathways that leads to poor prognosis in women with ER-positive disease, (2) blockade of JAK/STAT signaling, via JAK inhibition, in patients with activating IL-6 polymorphisms and/or upregulation of STAT3 tumor signaling will enhance the response to endocrine therapy, and (3) patients likely to respond to JAK inhibition can be identified by germline genotyping for IL-6 variants, and effectiveness of the targeted therapy will be measurable through tumor assessment of activated STAT signaling through upregulation of phospho- STAT3 and expression of STAT3 target genes.

We now propose a trial to determine whether addition of the JAK inhibitor, Ruxolitinib (INCB018424), enhances the activity of exemestane alone in women with ER-positive breast cancer who have relapsed after non-steroidal aromatase inhibitor and carry a germline polymorphism in IL-6, and to determine if tumor activation of STAT3 can identify patients most likely to respond to the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, invasive metastatic breast cancer.
* Estrogen-receptor positivity (defined by at least 5% staining by immunohistochemistry) on either the primary breast tumor or a metastatic biopsy.
* Postmenopausal status, defined as: either "surgical menopause" via oophorectomy, or "natural menopause" in which the patient has had no menses in the previous 12-month period. Premenopausal patients who have been been rendered amenorrheaic by tamoxifen must have a serum estradiol level <30 pg/ml after discontinuation of tamoxifen. Amenorrheaic premenopausal subjects must have a negative pregnancy test during screening (prior to enrollment) and must be advised to use adequate contraception throughout their participation.
* Prior therapy for the current malignancy: Patient must have 1) relapsed on or within 2 years of completing adjuvant hormonal therapy with a non-steroidal aromatase inhibitor, OR 2) failed a non-steroidal aromatase inhibitor in the metastatic setting. There is no limit to prior chemotherapy or hormonal regimens for this malignancy.
* At least one measureable lesion by RECIST or mainly lytic bone lesions in the absence of measurable disease. Bone-only disease is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function, defined as follows:

Bilirubin ≤ 1.5 x the upper limit of normal (ULN) Serum creatinine ≤ 1.5 x UNL or calculated creatinine clearance ≥ 60 mL/min, and

* For subjects without liver metastases: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
* For subjects with liver metastases: alanine aminotransferase (ALT) and aspartate aminotransferase ≤ 5 x ULN
* Adequate bone marrow function, defined as follows Absolute neutrophil count (ANC) >1500/mm3 Hemoglobin > 9 Platelets >100,000/mm3
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.

EXCLUSION CRITERIA:

* Chemotherapy, hormonal therapy or investigational anti-tumor therapy within 21 days of starting study treatment. Use of bone-building agents is allowed.
* Prior treatment with exemestane.
* Any type of investigational agent within 28 days before the first dose of study treatment.
* Unresolved clinically-meaningful toxicity due to prior therapy. Toxicity from previous treatment must be back to baseline or Grade ≤ 1, with the exception of neurotoxicity and alopecia.
* Untreated or uncontrolled brain metastases or evidence of leptomeningeal involvement of disease. Patients who have stable disease after radiotherapy for CNS disease are eligible. Testing for brain involvement in the absence of symptoms is not required as part of this protocol.
* Uncontrolled, intercurrent illness
* Known ongoing or active infection, including active hepatitis B or hepatitis C. Testing for hepatitis B or C is not required as part of this protocol.
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Symptomatic congestive heart failure, unstable angina pectoris, stroke or myocardial infarction within 3 months
* A baseline corrected QT interval (QTc) > 470 ms.
* The subject is known to be positive for the human immunodeficiency virus (HIV). Note: baseline HIV screening is not required
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela DiMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- First Stage: Ruxolitinib at 25 mg orally, twice daily and Exemestane, 25 mg orally once daily
  Ruxolitinib
  Exemestane
- Second Stage: Ruxolitinib at 15 mg orally, twice daily and Exemestane, 25 mg orally once daily
  Ruxolitinib
  Exemestane
Period: Overall Study
Arm/Group | First Stage | Second Stage
Started | 15 | 10
Completed | 15 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Stage | Second Stage | Total
Number analyzed (Participants) | 15 | 10 | 25
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 86] | 62 [51 to 83] | 60 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety will be assessed by evaluation of the number and severity adverse events as defined by the NCI CTCAE Version 4.0
Time Frame: 3 years
Population: 25 patients analyzed
Measure: Number; unit: participants
Arm/Group | First Stage | Second Stage
Number analyzed (Participants) | 15 | 10
participants | 5 | 1

2. Primary Outcome: Time to Progression
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Stage | Second Stage
Number analyzed (Participants) | 15 | 10
months | 2.8 [2.6 to 3.9] | 2.8 [2.6 to 3.9]

3. Secondary Outcome: Pharmacodynamic Assessment of Phospho-STAT3 Inhibition
Time Frame: 3 years
Measure: Median (Standard Deviation); unit: % inhibition of phosphorylated STAT3
Arm/Group | First Stage | Second Stage
Number analyzed (Participants) | 10 | 7
% inhibition of phosphorylated STAT3 | 24.5 (12.7) | 29 (26.4)

4. Secondary Outcome: Inflammatory Markers
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | First Stage | Second Stage
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/10
Other Adverse Events (participants affected / at risk) | 15/15 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Stage (N=15) | Second Stage (N=10)
neutropenic fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
elevated creatinine (Investigations) | 0 (0) | 1 (1)
hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Stage (N=15) | Second Stage (N=10)
anemia (grade 2) (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
neutropenia (grade 2) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
infection (grade 2) (Infections and infestations) | 1 (1) | 2 (2)
thrombocytopenia (grade 2) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
pain (grade 2) (General disorders) | 7 (7) | 8 (8)
psychiatric (grade 2) (Psychiatric disorders) | 4 (4) | 4 (4)
pulmonary (grade 2) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
nausea/vomiting (grade 2) (Gastrointestinal disorders) | 0 (0) | 2 (2)
other gastrointestinal (grade 2) (Gastrointestinal disorders) | 6 (6) | 3 (3)
elevated liver function test (grade 2) (Investigations) | 1 (1) | 1 (1)
pain (grade 1) (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8)
constipation (grade 1) (Gastrointestinal disorders) | 5 (5) | 2 (2)
fatigue (grade 2) (General disorders) | 4 (4) | 0 (0)
fatigue (grade 1) (General disorders) | 0 (0) | 4 (4)
fatigue (grade 3) (General disorders) | 0 (0) | 4 (4)
hypertension (grade 2) (Cardiac disorders) | 3 (3) | 1 (1)
hypertension (grade 3) (Cardiac disorders) | 1 (1) | 3 (3)
other gastrointestinal (grade 1) (Gastrointestinal disorders) | 3 (3) | 3 (3)
diarrhea (grade 1) (Gastrointestinal disorders) | 3 (3) | 0 (0)
diarrhea (grade 3) (Gastrointestinal disorders) | 0 (0) | 1 (1)
headache (grade 1) (Nervous system disorders) | 6 (6) | 1 (1)
headache (grade 2) (Nervous system disorders) | 1 (1) | 0 (0)
nausea/vomiting (grade 1) (Gastrointestinal disorders) | 3 (3) | 0 (0)
nausea/vomiting (grade 3) (Gastrointestinal disorders) | 0 (0) | 1 (1)
pain (grade 3) (General disorders) | 2 (2) | 1 (1)
anemia (grade 1) (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
anemia (grade 3) (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
pulmonary (grade 1) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8)
urinary (grade 1) (Renal and urinary disorders) | 3 (3) | 0 (0)
pulmonary (grade 3) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
elevated hepatic function (grade 1) (Investigations) | 8 (8) | 4 (4)
neutropenia (grade 1) (Investigations) | 3 (3) | 3 (3)
flu-like symptoms (grade 1) (Infections and infestations) | 5 (5) | 3 (3)
infection (grade 1) (Infections and infestations) | 3 (3) | 2 (2)
psychiatric (grade 1) (Psychiatric disorders) | 10 (10) | 2 (2)
neurological (grade 1) (Nervous system disorders) | 4 (4) | 2 (2)
hyponatremia (grade 1) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
dizziness (grade 2) (Nervous system disorders) | 1 (1) | 1 (1)
edema (grade 1) (General disorders) | 1 (1) | 0 (0)
edema (grade 2) (General disorders) | 2 (2) | 0 (0)
hyponatremia (grade 3) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
psychiatric (grade 3) (Psychiatric disorders) | 3 (3) | 0 (0)
psychiatric (grade 2) (Psychiatric disorders) | 3 (3) | 0 (0)
palpitations (grade 1) (Cardiac disorders) | 1 (1) | 0 (0)
pericarditis (grade 2) (Cardiac disorders) | 1 (1) | 0 (0)
decreased white blood cells (grade 1) (Investigations) | 4 (4) | 1 (1)
decreased white blood cells (grade 2) (Investigations) | 2 (2) | 2 (2)
vaginal bleeding (grade 1) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
premature menopause (grade 3) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
hot flashes (grade 1) (Vascular disorders) | 3 (3) | 1 (1)
hot flashes (grade 2) (Vascular disorders) | 1 (1) | 0 (0)
elevated creatinine (grade 1) (Renal and urinary disorders) | 2 (2) | 1 (1)
arthritis (grade 1) (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
dehydration (grade 1) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
pruritis (grade 1) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
blurred vision (grade 2) (Eye disorders) | 1 (1) | 0 (0)
urinary incontinence (grade 3) (Renal and urinary disorders) | 1 (1) | 0 (0)
urinary tract infection (grade 2) (Renal and urinary disorders) | 1 (1) | 0 (0)
neutropenia (grade 3) (Investigations) | 3 (3) | 0 (0)
decreased white blood cells (grade 3) (Investigations) | 3 (3) | 0 (0)
hypercalcemia (grade 2) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypermagnesemia (grade 1) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
type 2 diabetes (grade 2) (Endocrine disorders) | 1 (1) | 0 (0)
hypokalemia (grade 1) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
presyncope (grade 2) (Cardiac disorders) | 1 (1) | 0 (0)
decreased chloride (grade 1) (Investigations) | 0 (0) | 1 (1)
osteoporosis (grade 2) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
osteoporosis (grade 1) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
hypothyroidism (grade 2) (Endocrine disorders) | 3 (3) | 0 (0)
hypothyroidism (grade 1) (Endocrine disorders) | 1 (1) | 0 (0)
flu-like symptoms (grade 2) (Infections and infestations) | 0 (0) | 1 (1)
fracture (grade 2) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
leg cramps (grade 1) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
chest pressure (grade 1) (General disorders) | 1 (1) | 0 (0)
decreased AST (grade 2) (Investigations) | 0 (0) | 1 (1)
hypoalbuminemia (grade 2) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
fall (grade 2) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
elevated BNP (grade 1) (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes